CLINICAL TRIAL: NCT03508609
Title: An Open-Label Exploratory Clinical Study to Evaluate the Safety and Potential Bioactivity of CLBS16 in Patients With Coronary Microvascular Dysfunction (CMD) and Without Obstructive Coronary Artery Disease
Brief Title: Safety and Potential Bioactivity of CLBS16 in Patients With Coronary Microvascular Dysfunction and Without Obstructive Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cedars-Sinai Medical Center (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBS16-P01; 1R44HL135889-01 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-11

CONDITIONS: Coronary Microvascular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous CD34 cells (Experimental): Open label active treatment arm. Subjects receive autologous CD34 cells.
  Interventions: Biological: CLBS16

INTERVENTIONS:
Biological: CLBS16 — GCSF-mobilized autologous CD34 cells

SUMMARY:
This clinical trial will explore the safety and effect of GCSF-mobilized autologous ex vivo selected CD34 cells for the treatment of CMD in adults currently experiencing angina and with no obstructive coronary artery disease. Eligible subjects will receive a single intracoronary infusion of CLBS16.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥18
* History of and currently experiencing angina at least 3 times per week
* No obstructive coronary artery disease
* On stable medical therapy for 30 days prior to enrollment
* Must agree to use a reliable and acceptable method of contraception for the duration of participation
* Written informed consent

Exclusion Criteria:

* Myocardial infarction within 90 days
* Prior evidence of obstructive heart disease including PCI or CABG (or planned PCI or CABG)
* Diagnosis of other specific cardiac disease
* Must meet LVEF and GFR requirements
* Current use of coumadin or DOACs
* Hypersensitivity to G-CSF, apheresis or study product components
* Positive for HIV, hepatitis B or hepatitis C
* Active inflammatory or autoimmune disease, or chronic immunosuppressive state
* Drug abuse
* Pregnant or lactating
* Malignant neoplasm within 5 years
* History of Sickle Cell Disease
* Participation in another clinical study within 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Losordo, MD, Study Director — Chief Medical Officer
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henry TD, Bairey Merz CN, Wei J, Corban MT, Quesada O, Joung S, Kotynski CL, Wang J, Lewis M, Schumacher AM, Bartel RL, Takagi H, Shah V, Lee A, Sietsema WK, Losordo DW, Lerman A. Autologous CD34+ Stem Cell Therapy Increases Coronary Flow Reserve and Reduces Angina in Patients With Coronary Microvascular Dysfunction. Circ Cardiovasc Interv. 2022 Feb;15(2):e010802. doi: 10.1161/CIRCINTERVENTIONS.121.010802. Epub 2022 Jan 23. PMID 35067072
- [Derived] Rai B, Shukla J, Henry TD, Quesada O. Angiogenic CD34 Stem Cell Therapy in Coronary Microvascular Repair-A Systematic Review. Cells. 2021 May 8;10(5):1137. doi: 10.3390/cells10051137. PMID 34066713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous CD34 Cells
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Weight [Mean (Standard Deviation); unit: kg] | 83.36 (23.377)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.52 (7.322)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Coronary Flow Reserve
Description: Coronary Flow Reserve (CFR) is a measure of coronary microvascular function.
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
ratio | 0.62 (0.835)

2. Secondary Outcome: Change From Baseline in Microvascular Function as Assessed by Intracoronary Administration of Acetylcholine
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: % change in peak coronary blood flow
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
% change in peak coronary blood flow | 9.4 (105.408)

3. Secondary Outcome: Change From Baseline in Peripheral Arterial Tonometry
Time Frame: Day 180
Measure: Mean (Standard Deviation); unit: Reactive Hyperemia Index (ratio)
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
Reactive Hyperemia Index (ratio) | -0.19 (0.990)

4. Secondary Outcome: Change in Angina Frequency From Baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: angina episodes per day
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
angina episodes per day | -2.34 (2.938)

5. Secondary Outcome: Canadian Cardiovascular Society Angina Class
Description: Canadian Cardiovascular Society angina class grading scale is assessed according to the following scores:
  Grade 1: Ordinary physical activity does not cause angina, such as walking and climbing stairs. Angina with strenuous or rapid or prolonged exertion at work or recreation Grade 2: Slight limitation of ordinary activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, or in cold, or in wind, or under emotional stress, or only during the few hours after awakening. Walking more than two blocks on the level and climbing more than one flight of ordinary stairs at a normal pace and in normal conditions Grade 3: Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace Grade 4: Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest A higher grade is a worse outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: change in grade
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
change in grade | -1.21 (1.032)

6. Secondary Outcome: Change From Baseline in Seattle Angina Questionnaire
Description: The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: change in scale score
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
change in scale score
  Physical limitation scale | 16.81 (20.956)
  Angina stability scale | 23.61 (40.649)
  Angina frequency scale | 18.33 (28.952)
  Treatment satisfaction scale | 12.83 (19.925)
  Disease perception scale | 23.68 (24.417)

7. Secondary Outcome: Change From Baseline in SF-36 Scores
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: change in scale score
Arm/Group | Autologous CD34 Cells
Number analyzed (Participants) | 20
change in scale score
  Physical component scores | 6.66 (7.452)
  Mental component scores | 5.62 (8.628)
  Physical function | 5.94 (6.439)
  Role-physical | 9.81 (10.376)
  Bodily pain | 5.50 (6.681)
  General health | 3.53 (6.666)
  Vitality | 8.29 (8.666)
  Social functions | 7.91 (8.573)
  Role-emotional | 6.23 (11.287)
  Mental health | 4.13 (7.766)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were solicited from all subjects at each visit.
Arm/Group | Autologous CD34 Cells
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous CD34 Cells (N=20)
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Coronary artery dissection (Injury, poisoning and procedural complications) | 1
Ventricular fibrillation (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous CD34 Cells (N=20)
Bone Pain (Musculoskeletal and connective tissue disorders) | 11
Nausea (Gastrointestinal disorders) | 9
Headache (Nervous system disorders) | 6
Pain (General disorders) | 6
Angina pectoris (Cardiac disorders) | 6
Dizziness (Nervous system disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Paraesthesia oral (Gastrointestinal disorders) | 4
Catheter site pain (Injury, poisoning and procedural complications) | 3
Hepatic enzyme increased (Hepatobiliary disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fatigue (Musculoskeletal and connective tissue disorders) | 2
Pyrexia (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03508609/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT03508609/SAP_001.pdf